CLINICAL TRIAL: NCT00253630
Title: A Phase II Study of Suberoylanilide Hydroxamic Acid (SAHA) in Indolent Non-Hodgkin's Lymphoma
Brief Title: Vorinostat in Treating Patients With Low-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02843; NCI-2012-02843 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-63; PHII-63 (Other: City of Hope Comprehensive Cancer Center); 6963 (Other: CTEP); N01CM17101 (NIH); P30CA033572 (NIH); U01CA062505 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Nodal Marginal Zone Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive vorinostat PO BID on days 1-14. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with relapsed or refractory indolent non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor activity of SAHA (vorinostat) as assessed by the objective response rate, time to progression and survival in subjects with advanced lymphoma.

II. To assess the toxicity profile of SAHA in this patient population. III. To perform correlative laboratory investigations to confirm modulation of chromatin acetylation as the biologic target and attempt to gain insight into the downstream molecular mechanisms involved in the induction of apoptosis mediated by SAHA.

OUTLINE:

Patients receive vorinostat orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed/refractory indolent Non-Hodgkin's lymphoma (Included in this category are relapsed/refractory follicular center lymphomas grade I, II, III, relapsed /refractory marginal zone B-cell lymphoma (nodal and extranodal), relapsed/refractory mantle cell lymphoma)
* Patients must have measurable disease by computed tomography (CT) scan. positron emission tomography (PET) scan evaluations are desirable but not mandatory, so that patients with negative PET scans but measurable disease by CT are eligible
* Patients may have had up to four prior chemotherapeutic regimens; steroids alone and local radiation do not count as regimens (radiotherapy must have been completed at least 14 days prior to starting SAHA); rituxan alone does not count as a regimen, however, Bexxar or Zevalin do; the most recent therapy must have failed to induce a complete response, or there must be disease progression or recurrence after the most recent therapy
* Patients may be enrolled who relapse after autologous stem cell transplant if they are at least three months after transplant, and after allogeneic transplant if they are at least six months post transplant; to be eligible after either type of transplant, patients must have achieved platelet counts greater than 100,000/mcL, and white blood cell (WBC) greater than 1,000/mcL at some point after their transplant, and should have no active related infections (i.e. fungal or viral); in the case of allogeneic transplant relapse, there should be no active acute graft versus host disease (GvHD) of any grade, and no chronic graft versus host disease other than mild skin, oral, or ocular GvHD not requiring systemic immunosuppression
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status #2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits; patients with elevation of unconjugated bilirubin alone, as in Gilbert's Disease, are eligible
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine up to and including 2 mg/dl
* Premenopausal women must have a negative serum pregnancy test prior to entry on this study; the effects of SAHA on the developing human fetus at the recommended therapeutic dose are unknown; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks, rituximab within three months (unless there is evidence of progression) or radiotherapy within 2 weeks or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded; this does not include use of steroids, which may continue until two days prior to enrollment; low dose chlorambucil should be stopped two weeks prior to beginning SAHA; valproic acid should be stopped at least two weeks prior to enrollment; nitrosoureas and mitomycin should be stopped 6 weeks prior to enrollment
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases are excluded from this clinical trial unless the metastases are controlled after therapy and have not been treated with steroids within the past two months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA
* There must be no plans for the patient to receive concurrent hormonal, biological or radiation therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with SAHA
* Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are ineligible
* Patients with other active malignancies are ineligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Popplewell, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Kirschbaum M, Frankel P, Popplewell L, Zain J, Delioukina M, Pullarkat V, Matsuoka D, Pulone B, Rotter AJ, Espinoza-Delgado I, Nademanee A, Forman SJ, Gandara D, Newman E. Phase II study of vorinostat for treatment of relapsed or refractory indolent non-Hodgkin's lymphoma and mantle cell lymphoma. J Clin Oncol. 2011 Mar 20;29(9):1198-203. doi: 10.1200/JCO.2010.32.1398. Epub 2011 Feb 7. PMID 21300924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vorinostat)
Started | 37
Completed | 35
Not Completed | 2
Not completed — ineligible | 2

BASELINE CHARACTERISTICS:
Population: Two enrolled patients were ineligible due to diffuse B-cell lymphoma at start of treatment. Treatment was changed for these ineligible patients (within 2 months of enrollment) before a response evaluation. These patients were removed and are not included in the analysis.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 64.5 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Radiological assessment by CT and/or PET scan after every three cycles (every 3 months). Response assessed by the standard Cheson criteria (Cheson et al, J Clin Oncol 17:1244, 1999). Complete Remission (CR) - (a) FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative (b) Variably FDG-avid or PET negative; regression to normal size on CT; Partial Remission (PR) - 50% or greater decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT. Response Rate = CR + PR.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 35
percentage of participants | 29 [15 to 46]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Grades 3 & 4 adverse events definitely, probably or possibly related to treatment, graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 35
Participants
  ANC | 6
  Anorexia | 1
  Fatigue | 3
  Hemoglobin | 4
  Hypokalemia | 1
  Hyponatremia | 1
  Hypophosphatemia | 2
  Infection -Skin (cellulitis) | 1
  INR | 2
  Leukocytes (total WBC) | 4
  Lymphopenia | 5
  Myalgia | 1
  Mucositis/stomatitis | 1
  Platelets | 10
  Thrombosis/thrombus/embolism | 2

3. Secondary Outcome: Change in Histone Acetylation by Immunohistochemistry (IHC)
Description: Histone acetylation by IHC will be scored as -, +, ++, or +++, reflecting both the intensity of staining as well as the number of cells stained. Analysis will be descriptive, with the goal of describing baseline distributions and estimating the frequency and degree of changes from baseline.
Time Frame: Baseline to up to day 14
Population: Immunohistochemistry data was not collected and is not available for analysis.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Histone Acetylation by Western Blot (WB)
Description: Histone acetylation by WB will be recorded as the ratio of acetylated histone (measured by photodensitometry) divided by the total histone (H3 or H4), in order to control for the amount of protein loaded. Analysis will be descriptive, with the goal of describing baseline distributions and estimating the frequency and degree of changes from baseline.
Time Frame: Baseline to up to day 14
Population: Western Blot data was not collected and is not available for analysis.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

5. Secondary Outcome: 2-Year Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until Death from any cause, up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 35
percentage of participants | 77 [64 to 92]

6. Secondary Outcome: 2-Year Progression Free-Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression defined as any new lesion or increase by greater than 50% of previously involved sites from nadir.
Time Frame: Until death or progression, up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 35
percentage of participants | 37 [24 to 57]

ADVERSE EVENTS:
Time Frame: All adverse events were collected over a period of 10 years, 8 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Vorinostat)
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=35)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vorinostat) (N=35)
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Agitation (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 25
Anxiety (Psychiatric disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 14
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bilirubin increased (Investigations) | 2
Bladder infection (Infections and infestations) | 2
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 4
Blood glucose increased (Metabolism and nutrition disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 3
Cardiac disorder (Cardiac disorders) | 2
Cardiac valve disease (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 9
Coagulopathy (Investigations) | 1
Confusion (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Creatinine increased (Investigations) | 20
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Depressed level of consciousness (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 30
Diplopia (Eye disorders) | 1
Dizziness (Nervous system disorders) | 16
Dry eye syndrome (Eye disorders) | 2
Dry mouth (Gastrointestinal disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 14
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Ear pain (Ear and labyrinth disorders) | 1
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 13
Erectile dysfunction (Reproductive system and breast disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 3
Eye disorder (Eye disorders) | 3
Fatigue (General disorders) | 34
Fever (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 5
Flu-like symptoms (General disorders) | 14
Gait abnormal (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 4
Gastrointestinal pain (Gastrointestinal disorders) | 1
General symptom (General disorders) | 2
Glomerular filtration rate decreased (Renal and urinary disorders) | 1
Headache (Nervous system disorders) | 12
Hematoma (Vascular disorders) | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 30
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhage (Vascular disorders) | 2
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 6
Hemorrhage urinary tract (Renal and urinary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 3
Hot flashes (Vascular disorders) | 1
Hyperbilirubinemia (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypercholesterolemia (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Hypotension (Vascular disorders) | 5
Infection (Infections and infestations) | 2
INR increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 5
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Joint disorder (Musculoskeletal and connective tissue disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 7
Kidney pain (Renal and urinary disorders) | 1
Laboratory test abnormal (Investigations) | 2
Leukocyte count decreased (Investigations) | 14
Leukopenia (Investigations) | 9
Lip infection (Infections and infestations) | 1
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 4
Lymphopenia (Investigations) | 8
Mucositis oral (Gastrointestinal disorders) | 6
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 26
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Neurological disorder NOS (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 17
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Pain (General disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Palpitations (Cardiac disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Platelet count decreased (Investigations) | 30
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3
Proctoscopy abnormal (Gastrointestinal disorders) | 1
Protein urine positive (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash desquamating (Skin and subcutaneous tissue disorders) | 7
Rectal hemorrhage (Gastrointestinal disorders) | 1
Reproductive tract disorder (Reproductive system and breast disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 7
Rhinitis infective (Infections and infestations) | 1
Serum albumin decreased (Metabolism and nutrition disorders) | 13
Serum calcium decreased (Metabolism and nutrition disorders) | 6
Serum calcium increased (Metabolism and nutrition disorders) | 3
Serum cholesterol increased (Investigations) | 1
Serum glucose decreased (Metabolism and nutrition disorders) | 8
Serum magnesium decreased (Metabolism and nutrition disorders) | 2
Serum magnesium increased (Metabolism and nutrition disorders) | 2
Serum phosphate decreased (Metabolism and nutrition disorders) | 16
Serum potassium decreased (Metabolism and nutrition disorders) | 5
Serum potassium increased (Metabolism and nutrition disorders) | 3
Serum sodium decreased (Metabolism and nutrition disorders) | 9
Serum sodium increased (Metabolism and nutrition disorders) | 1
Serum triglycerides increased (Metabolism and nutrition disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Small intestinal mucositis (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 11
Sweating (Skin and subcutaneous tissue disorders) | 4
Taste alteration (Nervous system disorders) | 15
Thrombosis (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tremor (Nervous system disorders) | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper respiratory infection (Infections and infestations) | 4
Urinary frequency (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Vascular disorder (Vascular disorders) | 1
Vision blurred (Eye disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Vulvitis (Infections and infestations) | 1
Weight gain (Investigations) | 4
Weight loss (Investigations) | 12
Wound dehiscence (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Two enrolled patients were ineligible due to diffuse B-cell lymphoma at start of treatment. Their treatment was changed (within 2 months of enrollment) before a response evaluation. These patients were removed and are not included in the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less